CLINICAL TRIAL: NCT06464185
Title: A Prospective Clinical Study of CD3-CD20 Bisspecific Antibody Based Therapy Combined With CD19-CAR T Cells in the Treatment of Relapsed Refractory B-cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024021
Record Dates: First submitted 2024-05-21; First posted 2024-06-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: B-cell Non-Hodgkin Lymphoma
Keywords: Glofitamab; CAR-T; obinutuzumab
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bispecific antibody-based therapy combined with CAR-T cell therapy (Experimental)
  Interventions: Drug: Bispecific antibody-based combined with CAR-T cell therapy

INTERVENTIONS:
Drug: Bispecific antibody-based combined with CAR-T cell therapy — lymphocytes collection, and bispecific antibody-based therapy will be performed after successful Lymphocytes collection: Obinutuzumab:1000mg, cycle 1 day 1(C1D1) ,IV.
  Glofitamab: 2.5 mg, C1D8; 10 mg,C1D15 ; 30 mg,C2D1 and C3D1, IV. It can be combined with other Immunization therapy during the use of bispecific antibodies according to the patient's condition.
  On C4D1, the patient will be pretreated with fludarabine and cyclophosphamide (FC) regimen, and then infused with CART cells at a specific dose of 4 * 1000000/Kg. Bispecific antibody maintenance therapy will be initiated on month 1/2/3 after CART infusion. In Phase1 bispecific maintenance therapy will be divided into three dose groups, using a "3 + 3" dose escalation design. In Phase 2, bispecific maintenance therapy will be used at the MTD dose of Phase 1.

SUMMARY:
The aim of this study was to analyze the safety and efficacy of CD3-CD20 bispecific antibody-based therapy in combination with CD19-CAR-T cells for the treatment of relapsed and refractory B-cell Non-Hodgkin's （B-NHL） lymphoma.

The main questions it aims to answer：

1. The safety of CD3-CD20 bispecific antibody-based therapy in combination with CD19-CAR-T cells in B-NHL;
2. The effect of different doses of bispecific antibody maintenance therapy on CAR-T cell expansion.

DETAILED DESCRIPTION:
The study was divided into two phases:

In the previous phase Ib clinical study, the bispecific antibody was used for bridging therapy to reduce the Neoplasm load, followed by CART cell therapy. After CART cell therapy, low-dose bispecific antibody was used for maintenance, in order to explore the safe resistance of bispecific antibody combined with CAR-T cell therapy and further explore the effect of bispecific antibody combined with CAR-T cell therapy on CART cell expansion; Phase II study will expand the sample study to further clarify whether bispecific antibody combined with CAR-T cell therapy can further deepen the efficacy of CAR-T.

ELIGIBILITY:
Inclusion Criteria:

* The patient has fully understood the study and voluntarily signed the informed consent form (ICF)
* Must meet the diagnostic criteria for relapsed and refractory B-NHL and have evaluable disease lesions, in addition to the following characteristics for different types of B-NHL:

A, Diffuse large B-cell Lymphoma:

Patients with histologically confirmed DLBCL; Patients who must have received ,anthracyclines CD20 monoclonal antibodies and BTK inhibitors and other Drug therapy, and have received at least two lines of treatment and relapsed, not relieved or progressed within 24 months after the last line of treatment;

B, Relapsed and Refractory Follicular lymphoma (FL):

Tissue Biopsy proved FL: grade 1-3a; Must have received anthracyclines and CD20 monoclonal antibody Drug therapy, and have received at least two lines of treatment and relapsed, not remitted or progressed within 24 months after the last line of treatment;

C, Relapsed and Refractory Marginal zone lymphoma (MZL):

Histologically unequivocally confirmed MZL; Must have received anthracyclines and CD20 monoclonal antibody Drug therapy, and have received at least two lines of treatment and relapsed, not remitted or progressed within 24 months after the last line of treatment;

D, Relapsed and refractory Mantle cell lymphoma (MCL):

Histologically confirmed MCL; Relapsed or refractory after at least 2 lines of therapy (including anti-CD20 monoclonal antibody, anthracyclines or bendamustine, and BTKi);

E, Relapsed and refractory CLL:

Histologically confirmed CLL; Patients who have received at least Immunochemotherapy and have Drug therapy to both BTK inhibitors and BCL2 inhibitors Drug resistance;

F, Relapsed and refractory WM:

Patients with histologically confirmed WM; Patients who must have received anthracyclines, CD20 monoclonal antibodies and BTK inhibitors and other Drug therapy, and have received at least two lines of treatment and relapsed, not relieved or progressed within 24 months after the last line of treatment;

* ECOG score 0-1
* Laboratory test: Neutrophils 0.5 x 10 ^ 9/L; platelets 30 x 10 ^ 9/L; Bilirubin total 2 x upper limit; GPT/Glutamic-oxaloacetic transferase 3 x upper limit. Creatinine clearance ≥ 30 mL/min.
* The expected survival time of patients is ≥ 6 months;

Exclusion Criteria:

* Neoplasm malignant other than B-NHL (except active central nervous system lymphoma) diagnosed or treated within the past year; Patients who received anti Neoplasm therapy (including chemotherapy, targeted therapy, hormone therapy, traditional Chinese medicine with anti neoplasm activity, etc.) or participated in other clinical trials and received the investigational drug within 4 weeks before the first use of the investigational drug;
* Liver renal impairment not related to lymphoma: GPT (ALT) > 3 times the upper limit of normal, glutamic-oxaloacetic transferase (AST) > 3 times the upper limit of normal, bilirubin total (TBIL) > 2 times the upper limit of normal, serum creatinine clearance rate < 30ml/min;
* Other serious medical diseases that will affect the study (such as uncontrolled Diabetes mellitus, gastric ulcer, other serious heart lung disease, etc.), and the right to decide belongs to the investigator.
* Cardiac function and disease meet one of the following conditions:

A, Long QTc syndrome or QTc interval > 480 MS; B, Complete left bundle branch block, grade II or III AV block; C, Serious, uncontrolled arrhythmia requiring drug therapy; D, New York Heart Association Heart disorder grade ≥ III; E, Cardiac Ejection Fraction (LVEF) less than 50%; F, Ischaemia, unstable Angina pectoris, history of severe unstable Ventricular arrhythmia or any other Arrhythmia requiring treatment, history of clinically significant Pericardial disease, or Electrocardiogram evidence of acute Myocardial infarction or active conduction system abnormalities within 6 months prior to recruitment;

* Known history of Infection human Immunodeficiency virus (HIV) or active Hepatitis B virus (HBV) Infection, or any uncontrolled active Injection requiring intravenous Systemic infection of antibiotics; Patients in the past 14 days received a large surgery (excluding lymph node Biopsy) or expected treatment in the need for a large Surgery;
* Previous or current other neoplasm malignant (except effectively controlled skin Basal cell carcinoma without melanoma, breast/In situ cancer of cervix, and other effectively controlled Neoplasm malignant without treatment within the past five years
* Pregnancy or lactating women, women of childbearing age who did not take contraception measures;
* Hypersensitivity to the drugs or ingredients used;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and severity of adverse events (AE) of patients treated with bispecific antibody combined with CD19-CAR-T cells in B-NHL.（Assessed by CTCAE criteria v5 and ASTCT 2019 criteria for CRS/ICANS adverse events.） | Up to 30 days after last treatment.From registration and during the bridging treatment, until end of post-treatment safety reporting window (up to six months after last dose of glofitamab)
  Assess the safety and toxicity of CD3-CD20 bispecific antibody-based therapy in combination with CD19-CAR-T cells in B-NHL. Assessed in all patients given at least one dose of study treatment and infused.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | Up to 12 months after last treatment
Overall Response Rate (ORR) | Up to 12 months after last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China